CLINICAL TRIAL: NCT01063855
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study of the Efficacy and Safety of Dapoxetine in Men With Premature Ejaculation and Concomitant Erectile Dysfunction Treated With a Phosphodiesterase-5 Inhibitor
Brief Title: Concomitant Use of PriLigy in Men Treated for Erectile Dysfunction
Acronym: COUPLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016486; R096769PRE3008 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2009-013616-12 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction
Keywords: Erectile Dysfunction; Sexual Dysfunction; Dapoxetine hydrochloride; PRILIGY; Premature ejaculation; Serotonin Uptake Inhibitors; Sildenafil (Viagra); Vardenafil (Levitra); Tadalafil (Cialis)
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological; Premature Ejaculation | interventions — dapoxetine; Phosphodiesterase 5 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapoxetine + PDE5I (Experimental): Dapoxetine 30 mg to 60 mg tablets 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + a PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction.
  Interventions: Drug: Dapoxetine; Drug: PDE5I (phosphodiesterase-5 inhibitor)
- Placebo + PDE5I (Placebo Comparator): Placebo tablets identical in appearance to dapoxetine taken 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + a PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction.
  Interventions: Drug: Placebo; Drug: PDE5I (phosphodiesterase-5 inhibitor)

INTERVENTIONS:
Drug: Placebo — Tablets identical in appearance to dapoxetine taken 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks.
  Arms: Placebo + PDE5I
Drug: Dapoxetine — 30 mg to 60 mg tablets 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks.
  Arms: Dapoxetine + PDE5I
Drug: PDE5I (phosphodiesterase-5 inhibitor) — Patients were to be using a stable regimen of a PDE5-I (i.e., sildenafil, vardenafil, or tadalafil), as reported by the patient for the treatment of erectile dysfunction (ED) for at least 3 months before screening and up to 12 weeks during treatment in the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dapoxetine compared to placebo in men with premature ejaculation and erectile dysfunction who are currently being treated with a phosphodiesterase-5 inhibitor (ie, sildenafil, vardenafil, or tadalafil) for erectile dysfunction.

DETAILED DESCRIPTION:
Premature ejaculation (PE) and erectile dysfunction (ED) are forms of sexual dysfunction in men. An objective measurement of PE in clinical studies is the intravaginal ejaculatory latency time (IELT), which is the time it takes for a man to ejaculate during sexual intercourse (as measured by stopwatch). This is a multicenter, double-blind (neither the physician or the study participant will know the identity of the treatment assigned), randomized (study drug assigned by chance) efficacy and safety study of dapoxetine compared with placebo (a sugar pill) in men with premature ejaculation who are currently being treated for ED with a phosphodiesterase 5 (PDE-5) inhibitor such as sildenafil, vardenafil, or tadalafil. A maximum of 656 men 18 years or older (hereafter referred to as study participants) who have received treatment with a PDE-5 inhibitor for at least 3 months prior to study entry will be enrolled. The study will last approximately 18 weeks and includes a 4-week screening period, a 12-week treatment period, and a follow-up telephone contact approximately 2 weeks after the end of treatment. Both the study participant and his partner will be required to attend the screening visit and to sign an informed consent form documenting that they understand and agree to the requirements for the study. After initial screening procedures are completed, study participants who qualify for the study will enter a 4-week screening period. During the 4 weeks, the study participant and his partner will be provided with a stopwatch to time and record the IELT during all attempts at sexual intercourse. At the next scheduled clinic visit which is Day 1 of the double-blind treatment period, study participants who continue to qualify for the study will be assigned by chance (like flipping a coin) to receive 1 of 2 study treatments (dapoxetine or placebo) for 12 weeks in addition to prescribed treatment with a PDE-5 inhibitor. Study participants will be instructed to take study drug with or without food with at least 1 full glass of water approximately 1 to 3 hours before sexual activity (no more than 1 dose should be taken within a 24-hour period). During the 12-week treatment period, the study participant and his partner will be asked to time and record the IELT during all attempts at sexual intercourse on Treatment Event Logs provided. Study participants will return to the clinic after 4, 8 and 12 weeks of treatment for routine safety assessments (including review of Treatment Event Logs returned) and to be dispensed study drug. Following 12 weeks of treatment (or at the time of early withdrawal from the study) end-of-treatment safety and efficacy evaluations will be performed at the final clinic visit. Approximately 2 weeks later, a follow up telephone call will be made to the study participant to collect information on any adverse events that may have occurred or concomitant therapy received since the time of the last clinic visit. The primary outcome measure in the study is the average IELT, as measured by stopwatch, during sexual intercourse at the end of the treatment period (Week 12). Safety will be monitored during the study by evaluating adverse events, physical examination findings, results from clinical laboratory tests, and concomitant medication usage. An Independent Data Monitoring Committee (IDMC) will be established to monitor the safety and efficacy of study participants during the study. In addition, an interim (preliminary) analysis will be performed during the study to monitor safety and efficacy after approximately 268 men have completed 12 weeks of treatment (also includes any study participants who did not complete treatment and were withdrawn early from the study). Study participants will receive either dapoxetine or matching placebo tablets at a dose of 30 mg prn (as needed) taken orally (by mouth) with or without food with at least 1 full glass of water approximately 1 to 3 hours before sexual activity (not to be taken more than once every 24 hours). At Weeks 4 or 8, the dose of dapoxetine or matching placebo may be increased to a maximum of 60 mg prn if specific predefined criteria are met or be subsequently decreased from 60 to 30 mg at Weeks 4 or 8.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of erectile dysfunction (ED), International Index of Erectile Function (IIEF) score >=21 at screening and baseline, and receiving treatment with a stable regimen of a phosphodiesterase 5 (PDE 5) inhibitor (ie, sildenafil, vardenafil, or tadalafil) for the treatment of ED for at least 3 months before screening
* Study participant in a stable, monogamous sexual relationship with the same woman for at least 6 months before screening and plan to maintain this relationship for the duration of the study
* Study participant medically stable (ie, in good general health) on the basis of physical examination, medical history, vital signs, 12 lead ECG, and clinical laboratory tests performed at screening

Exclusion Criteria:

* History suggestive of syncope (a condition characterized by a loss of consciousness)
* History of medical events such as surgical interventions or neurologic conditions (eg, multiple sclerosis), trauma, or infections that are associated with the development of symptoms of premature ejaculation (PE) and considered a potential cause of PE
* Current major psychiatric disorder such as mood disorder, anxiety disorder, schizophrenia, mania, suicidal ideation, other psychotic disorder, or alcoholism
* Known allergy, hypersensitivity, or intolerance to selective serotonin reuptake inhibitors (SSRIs) or selective noradrenaline reuptake inhibitors (SNRIs)
* Taken another investigational drug (or vaccine) within 30 days or used an investigational medical device within 6 months before screening, or enrolled in another investigational study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (69):
- United States (19):
  - Decatur, Alabama
  - Huntsville, Alabama
  - Englewood, Colorado
  - Aventura, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - West Palm Beach, Florida
  - Evansville, Indiana
  - Fort Wayne, Indiana
  - Baltimore, Maryland
  - Olive Branch, Mississippi
  - Kansas City, Missouri
  - Poughkeepsie, New York
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Salem, Oregon
  - Ettrick, Virginia
  - Middleton, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Ciudad Autonoma de
- Australia (4):
  - Malvern
  - Maroubra
  - Perth
  - St Leonards
- Belgium (3):
  - Brussels
  - Edegem
  - Liège
- Canada (8):
  - Coquitlam, British Columbia
  - Guelph, Ontario
  - Newmarket, Ontario
  - Oakville, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
- France (7):
  - Garches
  - Lille
  - Lyon
  - Marseille
  - Nîmes
  - Paris
  - Toulouse
- Malaysia (3):
  - Kuala Lumpur
  - Kuching
  - Petaling Jaya
- Mexico (4):
  - Cd. de Mexico
  - Culiacán
  - Durango
  - Monterrey
- Poland (5):
  - Katowice
  - Lodz
  - Lublin
  - Szcezecin
  - Wroclaw
- Russia (3):
  - Moscow
  - Saint Peterburg
  - Saint Petersburg
- South Korea (4):
  - Chunjoo
  - Kwangjoo
  - Pusan
  - Seoul
- Taiwan (2):
  - Kaohsiung City
  - Taoyuan District
- United Kingdom (5):
  - Chipping Norton
  - Leeds Yorkshire
  - Lichfield
  - Reading
  - South Brent

REFERENCES:
- [Derived] McMahon CG, Giuliano F, Dean J, Hellstrom WJ, Bull S, Tesfaye F, Sharma O, Rivas DA, Aquilina JW. Efficacy and safety of dapoxetine in men with premature ejaculation and concomitant erectile dysfunction treated with a phosphodiesterase type 5 inhibitor: randomized, placebo-controlled, phase III study. J Sex Med. 2013 Sep;10(9):2312-25. doi: 10.1111/jsm.12236. Epub 2013 Jul 11. PMID 23845016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study R096769-PRE-3008 was conducted at 69 study centers in 13 countries between 27 April 2010 and 31 August 2011.
Pre-assignment Details: Of the 495 randomized patients, 429 patients completed the study, and 66 patients were discontinued from the study. All randomized patients (N=495) were included in the intent-to-treat analysis set of patients for efficacy and safety.
Groups:
- PDE5I + PLACEBO: Placebo tablets identical in appearance to dapoxetine taken 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction.
- PDE5I + DPX: Dapoxetine 30 mg to 60 mg tablets 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction.
Period: Overall Study
Arm/Group | PDE5I + PLACEBO | PDE5I + DPX
Started | 245 | 250
Completed | 208 | 221
Not Completed | 37 | 29
Not completed — Adverse Event | 4 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 8 | 4
Not completed — Pregnancy | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Reason not specified | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PDE5I + PLACEBO | PDE5I + DPX | Total
Number analyzed (Participants) | 245 | 250 | 495
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 228 | 231 | 459
  >=65 years | 17 | 19 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.96) | 49.5 (11.23) | 48.7 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 245 | 250 | 495
Baseline BMI [Mean (Standard Deviation); unit: kg/cm2] | 27.2 (4.50) | 27.1 (4.55) | 27.2 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: The Average Intravaginal Ejaculatory Latency Time (IELT) at Week 12
Description: The intravaginal ejaculatory latency time (IELT) is the time it takes for a man to ejaculate during sexual intercourse (as measured by stopwatch). The data below show the average IELT measured in minutes at Baseline (before treatment) to Endpoint (after 12 weeks of treatment). In this study, patients took placebo or dapoxetine along with a stable dose of a phosphodiesterase-5 inhibitor (PDE5I) prescribed prior to study entry for the treatment of erectile dysfunction.
Time Frame: Baseline, Week 12
Population: The intent-to-treat (ITT) analysis set included all randomized patients. Missing efficacy data at Week 12 was imputed based on the last postbaseline observation carried forward (LPOCF) method.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- PDE5I + Placebo (Baseline); PDE5I + Placebo (Week 12): Placebo tablets identical in appearance to dapoxetine taken 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction.
- PDE5I + Dapoxetine (Baseline); PDE5I + Dapoxetine (Week 12): Dapoxetine 30 mg to 60 mg tablets 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction
Arm/Group | PDE5I + Placebo (Baseline) | PDE5I + Placebo (Week 12) | PDE5I + Dapoxetine (Baseline) | PDE5I + Dapoxetine (Week 12)
Number analyzed (Participants) | 241 | 230 | 249 | 240
minutes | 1.1 (0.53) | 3.4 (3.54) | 1.1 (0.55) | 5.2 (5.78)
Statistical Analysis 1: Comparison: PDE5I + Placebo (Baseline) vs PDE5I + Placebo (Week 12) vs PDE5I + Dapoxetine (Baseline) vs PDE5I + Dapoxetine (Week 12); Null Hypothesis: No difference at Week 12 last postbaseline observations carried forward (LPOCF) Alternative Hypothesis:- Difference at Week 12 LPOCF >0; Test type: Superiority or Other; p < 0.001, ANCOVA — To properly adjust for multiplicity, a hierarchical (step-down) testing procedure with a priori ordered hypothesis was used to control the family-wise type I error was rate; ANCOVA model included treatment, PDE5I stratum, baseline Average IELT stratum, and region, as cofactors and baseline Average IELT as a covariate; Median Difference (Final Values) = 1.69, 95% CI 2-sided [0.837 to 2.542], Standard Error of Mean 0.430 — Estimates are based on two-stage sequential analysis using information fraction based weighted test statistics for PDE5I + Dapoxetine arm minus PDE5I + Placebo arm difference

2. Secondary Outcome: The Percentage of Patients Reporting At Least a 2-category Increase in Control Over Ejaculation
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's control over ejaculation on a 5-point scale from "Very poor, Poor, Fair, Good, to Very Good." The percentage of patients who reported at least a 2-category increase in control over ejaculation is provided in the table below.
Time Frame: At the end of treatment (Week 12)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Groups:
- PDE5I + Dapoxetine: Dapoxetine 30 mg to 60 mg tablets 1 to 3 hours before sexual activity prn (as needed) not to be taken more than once every 24 hours for 12 weeks + PDE5I (phosphodiesterase-5 inhibitor) prescribed prior to study entry for the treatment of erectile dysfunction.
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 229 | 246
Percentage of Patients | 32.3 | 45.9
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; Null hypothesis: No difference at Week 12 last postbaseline observation carried forward (LPOCF). Alternative hypothesis: Difference at Week 12 LPOCF > 0; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — A hierarchical (step-down) testing procedure with a priori ordered hypothesis was used to control the family-wise type 1 error rate; Cochran-Mantel-Haenszel (CMH) test, controlling for type of PDE5I stratum, baseline average IELT stratum, and region; Risk Difference (RD) = 13.6, 95% CI 2-sided [4.9 to 22.3] — Risk Difference (RD) = PDE5I + Dapoxetine arm - PDE5I + placebo arm

3. Secondary Outcome: The Percentage of Patients Who Achieved 1-category or Greater Decrease (Improvement) in Personal Distress Related to Ejaculation
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of distress related to the speed of ejaculation on a 5-point scale from "Very poor, Poor, Fair, Good, to Very Good." The percentage of patients who achieved 1-category or greater decrease (improvement) in personal distress related to the speed of ejaculation is provided in the table below.
Time Frame: At Endpoint (After 12 weeks of treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 229 | 246
Percentage of Patients | 67.2 | 76.4
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; Null Hypothesis: No difference at Week 12 last postbaseline observation carried forward (LPOCF); Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; The Cochran-Mantel-Haenszel (CMH) test, controlling for type of PDE5I stratum, baseline average IELT stratum, and region; Risk Difference (RD) = 9.2, 95% CI 2-sided [1.1 to 17.2] — Risk Difference (RD) = PDE5I + Dapoxetine arm - PDE5I + Placebo arm

4. Secondary Outcome: The Percentage of Patients Reporting a Composite Score of At Least a 2-category Increase in Control Over Ejaculation and At Least a 1-category Decrease in Personal Distress
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of distress related to the speed of ejaculation and control over ejaculation on a 5-point scale from "Very poor, Poor, Fair, Good, to Very Good." The percentage of patients who reported a composite score of at least a 2-category increase in control over ejaculation and at least a 1-category decrease (improvement) in personal distress is provided in the table below.
Time Frame: At the end of treatment (Week 12)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 229 | 246
Percentage of Patients | 30.6 | 43.5
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; Null Hypothesis: No difference at Week 12 last postbaseline observation carried forward (LPOCF) Alternative Hypothesis: PDE5I + Dapoxetine is superior to PDE5I + Placebo with respect to the outcome measure at Week 12 LPOCF; Test type: Superiority or Other; p = 0.002, Regression, Logistic — To properly adjust for multiplicity, a hierarchical (step-down) testing procedure with a priori ordered hypothesis was used to control the family-wise type I error; Logistic Regression model included treatment, type of PDE5i stratum, baseline Average IELT stratum, and region, as factors; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.204 to 2.619] — Estimates are based on two-stage sequential analysis using information fraction based weighted test statistics for PDE5I + Dapoxetine arm over PDE5I + Placebo arm ratio

5. Secondary Outcome: The Percentage of Patients Who Achieved a 1-category or Greater Increase in Satisfaction With Sexual Intercourse
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of satisfaction with intercourse on a 5-point scale from "Very poor, Poor, Fair, Good, to Very Good." The percentage of patients who achieved 1-category or greater increase in satisfaction with sexual intercourse is provided in the table below.
Time Frame: Endpoint (After 12 weeks of treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 229 | 246
Percentage of Patients | 55.0 | 66.3
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; Null Hypothesis: No difference at Week 12 last postbaseline observation carrried forward (LPOCF) Alternative Hypothesis:- PDE5I + Dapoxetine is superior to PDE5I + Placebo with respect to the outcome measure at Week 12 LPOCF; Test type: Superiority or Other; p = 0.007, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.108 to 2.394] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: The Percentage of Patients Reporting At Least a "Better" Response to Treatment
Description: The "Clinical Global Impression of Change" (CGIC) was used to assess the degree of improvement the patient experienced with premature ejaculation (PE) since initiating treatment with study drug on a 7-point scale from "Much worse, Worse, Slightly worse, No change, Slightly better, Better, to Much better". The percentage of patients who reported improvement in PE of at least "better" at Endpoint (after 12 weeks of treatment) is provided in the table below.
Time Frame: Endpoint (After 12 weeks of treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 229 | 246
Percentage of Patients | 35.4 | 56.5
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; Null Hypothesis: No difference at Week 12 last postbaseline observation carried forward (LPOCF) Alternative Hypothesis:- PDE5I + Dapoxetine is superior to PDE5I + Placebo with respect to the outcome measure at Week 12; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.642 to 3.568] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: The Percentage of Patients Who Reported At Least a 1-category Decrease (Improvement) in Interpersonal Difficulty Related to Ejaculation
Description: The Premature Ejaculation Profile (PEP), a patient-reported outcome measure was used to rate the patient's level of interpersonal difficulty related to ejaculation on a 5-point scale from "Very poor, Poor, Fair, Good, to Very Good." The percentage of patients who reported at least a 1-category decrease (improvement) in interpersonal difficulty related to ejaculation is provided in the table below.
Time Frame: Endpoint (After 12 weeks of treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 229 | 246
Percentage of Patients | 61.6 | 67.5
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; Null Hypothesis: No difference at Week 12 last postbaseline observation carried forward (LPOCF) Alternative Hypothesis:- PDE5I + Dapoxetine is superior to PDE5I + Placebo with respect to the outcome measure at Week 12 LPOCF; Test type: Superiority or Other; p > 0.05, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.897 to 1.965] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: The Percentage of Patients Reporting At Least a "Slightly Better" Response to Treatment
Description: The "Clinical Global Impression of Change" (CGIC) was used to assess the degree of improvement the patient experienced with premature ejaculation (PE) since initiating treatment with study drug on a 7-point scale from "Much worse, Worse, Slightly worse, No change, Slightly better, Better, to Much better". The percentage of patients who reported improvement in PE of at least "slightly better" at Endpoint (after 12 weeks of treatment) is provided in the table below.
Time Frame: Endpoint (After 12 weeks of treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | PDE5I + Placebo | PDE5I + Dapoxetine
Number analyzed (Participants) | 230 | 240
Percentage of Patients | 66.9 | 91.3
Statistical Analysis 1: Comparison: PDE5I + Placebo vs PDE5I + Dapoxetine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.425 to 3.423] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 18 weeks.
Arm/Group | PDE5I + PLACEBO | PDE5I + DPX
Serious Adverse Events (participants affected / at risk) | 4/245 | 3/250
Other Adverse Events (participants affected / at risk) | 45/245 | 73/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PDE5I + PLACEBO (N=245) | PDE5I + DPX (N=250)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 1
Miscarriage of Partner (Social circumstances) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PDE5I + PLACEBO (N=245) | PDE5I + DPX (N=250)
Palpitations (Cardiac disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 4
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Eye Pain (Eye disorders) | 0 | 1
Eyelid Ptosis (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 9
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 23
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Adverse Drug Reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Irritability (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bacterial Food Poisoning (Infections and infestations) | 0 | 1
Ear Infection Viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3
Oral Herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1
Back Injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint Sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1
Gastric Ph Decreased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 6
Dizziness Exertional (Nervous system disorders) | 1 | 0
Dizziness Postural (Nervous system disorders) | 1 | 6
Headache (Nervous system disorders) | 12 | 11
Lethargy (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Euphoric Mood (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal Cyst (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0
Penis Disorder (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days